CLINICAL TRIAL: NCT04113564
Title: A Randomized, Open-label, Single-dose, 2-way Crossover Study to Compare the Relative Bioavailability of Orally Administered Remimazolam to an Intravenous Formulation in Healthy Volunteers
Brief Title: Absolute Oral Bioavailability of Remimazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CNS7056-016
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Bioavailability
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV remimazolam (Experimental): IV remimazolam administration of 0.025 mg/kg body weight
  Interventions: Drug: Remimazolam
- Oral remimazolam (Experimental): Oral remimazolam Administration of 0.14 mg/kg Body weight
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam
  Other Names: CNS7056

SUMMARY:
A randomized, open-label, single-dose, 2-way crossover study to compare the relative bioavailability of orally administered remimazolam to an intravenous formulation in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study, willing to give written informed consent prior to the initiation of any protocol-specific procedures, and willing to comply with the study restrictions.
2. Had to be able to speak, read, and understand English sufficiently to allow completion of all study assessments.
3. Gender : males and/or females
4. Age : 18 - 55 years, inclusive
5. Body mass index (BMI) : 18.0 - 32.0 kg/m2
6. Weight : ≥50 kg
7. Healthy status was defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, clinical chemistry, serology, and urinalysis.
8. Ability and willingness to abstain from alcohol, caffeine, and xanthine-containing beverages or food (eg, coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) prior to admission to the clinical facility on Day -1 until study discharge.
9. All values for hematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Investigator.
10. Females of childbearing potential and males and their female partner(s) of childbearing potential had to agree to use 2 forms of contraception, 1 of which had to be a barrier method, during the study and for 90 days after the last drug administration. Acceptable barrier forms of contraception were condom and diaphragm. Acceptable non-barrier forms of contraception for this study were an intrauterine device (IUD) and/or spermicide.
11. For females: a negative pregnancy test at Screening and Day -1.
12. Postmenopausal females: defined as 12 months with no menses prior to Screening and a serum follicle stimulating hormone (FSH) >40 IU/L at Screening.
13. All non-regular medication (including over-the-counter [OTC] medication, health supplements, and herbal remedies such as St. John's Wort extract) must have been stopped at least 14 days prior to admission to the clinical research center. An exception was made for paracetamol (acetaminophen), which was allowed up to admission to the clinical research center.

Exclusion Criteria:

1. Women who were pregnant or lactating.
2. Males with female partners who were pregnant or lactating.
3. Use of any investigational drug or device within 30 days of the first dose of study medication.
4. Any disease which, in the opinion of the Investigator, posed an unacceptable risk to the subjects.
5. Known allergy, hypersensitivity or prior intolerance to benzodiazepine derivates or flumazenil, or a medical condition such that these agents were contraindicated.
6. The use of tobacco products within 60 days prior to the first drug administration.
7. Routine or chronic use of more than 3 grams of acetaminophen daily.
8. Strenuous activity, sunbathing and contact sports within 48 hours (2 days) prior to admission to the clinical facility and for the duration of the study.
9. History of donation of more than 450 mL of blood within 60 days prior to dosing in the clinical research center or planned donation before 30 days had elapsed since intake of study drug.
10. Plasma or platelet donation within 7 days of dosing and throughout the entire study.
11. History of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol). Alcohol consumption was prohibited from 48 hours prior to admission to the clinical facility and throughout the entire study until discharge.
12. Positive screening test for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, or anti-human immunodeficiency virus (HIV) 1 and 2 antibodies.
13. Positive results for drugs of abuse, including cotinine, in the urine at Screening or Day -1.
14. Positive results for alcohol abuse, as determined by alcohol breath test, at Screening or Day -1.
15. Inability to be venipunctured or tolerate venous access as determined by the Investigator or designee.
16. History of clinically significant, recent/current and nonremote suicidal ideations or suicide attempts that, in the opinion of the Investigator, posed an unacceptable risk to the subject for participating in the study.
17. Any major surgery within 4 weeks of study drug administration. NOTE: Any parameter/test could be repeated at the Investigator's discretion during Screening and/or on Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability of remimazolam | Day 1 (pre-dode) to Day 3
  Single-dose bioavailability of an oral formulation of remimazolam relative to an IV formulation of remimazolam in healthy male and female subjects

SECONDARY OUTCOMES:
Maximum Plasma concentration (Cmax) | Day 1 (pre-dode) to Day 3
  Maximum observed plasma concentration
Time to Maximum Plasma concentration (Tmax) | Day 1 (pre-dode) to Day 3
  Time to attain maximum observed plasma concentration
Area under the plasma concentration-time curve (AUC0-t) | Day 1 (pre-dode) to Day 3
  Area under the plasma concentration-time curve from time 0 up to the time of the last measurable concentration
Elimination half-life (T1/2) | Day 1 (pre-dode) to Day 3
  Terminal elimination half-life
Clearance (CL/F) | Day 1 (pre-dode) to Day 3
  Apparent oral clearance
Volume of Distribution (Vz/F) | Day 1 (pre-dode) to Day 3
  Apparent volume of distribution at terminal phase
Incidences of Treatment-emergent adverse events | Day 1 (pre-dode) to Day 3
  Incidences of Treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Searle, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA Health Sciences (PRA) - Early Development Services (EDS), Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pesic M, Stohr T, Ossig J, Borkett K, Donsbach M, Dao VA, Webster L, Schippers F. Remimazolam Has Low Oral Bioavailability and No Potential for Misuse in Drug-Facilitated Sexual Assaults, with or Without Alcohol: Results from Two Randomised Clinical Trials. Drugs R D. 2020 Sep;20(3):267-277. doi: 10.1007/s40268-020-00317-0. PMID 32757149